CLINICAL TRIAL: NCT01648010
Title: An Open Label Study Evaluating Short Term Safety and Tolerability of Patients With MUSCLE INVASIVE BLADDER CANCER- for Intravesical Instillation Mitomycin c Mixed With Disposable Device Which Prevents Drug Drainage Out of the Patient's Bladder
Brief Title: Safety and Tolerability Study Which Evaluate Intravesical Instillation With Mitomycin C Mixed With TC-3 Drug Retaining Hydrogel Device In Patients With Muscle Invasive Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: TAS-4M-PR-H-127-1; HTA 5972 (Other: Israeli Ministry of Health)
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2012-12

CONDITIONS: Carcinoma of Urinary Bladder, Invasive
Keywords: Non Muscle Invasive Bladder Cancer; Carcinoma of urinary bladder, invasive; Intravesical instillation; Mitomycin C; Hydrogel; Reverse thermal gelation; Drug retention; radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TC-3 gel (Experimental): TC-3 gel group undergo intravesical instillation of the investigatory device
  Interventions: Device: TC-3 gel
- MMC- gel (Experimental): MMC gel group undergo intravesical instillation of the reverse thermal gelation device mixed with MMC
  Interventions: Device: TC-3 gel mixed with Mitomycin C (MMC)

INTERVENTIONS:
Device: TC-3 gel — One intravesical instillation of 40 cc of TC-3 hydrogel is instilled using catheter.
  Arms: TC-3 gel
Device: TC-3 gel mixed with Mitomycin C (MMC) — One intravesical instillation of 40 cc of TC-3 gel mixed with 40 mg MMC will be instilled using catheter
  Other Names: MMC Gel
  Arms: MMC- gel

SUMMARY:
The purpose of this study is to evaluate the safety of intravesical instillation of TC-3 Hydrogel disposable device for retention of mitomycin C chemotherapeutic drug in the urinary bladder.

DETAILED DESCRIPTION:
Non-muscle-Invasive Bladder cancer is mainly treated by tumor resection (Trans Urethral Resection - TUR), followed by series of intravesical instillations of prophylactic chemotherapeutic drugs as Mitomycin C (MMC).This treatment approach is limited due to rapid dilution the chemotheraputic drug by the incoming urine and clearance by urination.

TheraCoat core technology is based on a reverse thermal (low viscosity at 5°C) degradable gel (TC-3)for MMC retention in the urinary bladder.

Prior to instillation, the TC-3 hydrogel,in a liquid state, is mixed with MMC.TC-3 mixed with MMC is instilled to the bladder by a catheter.Following gel insertion to the bladder, the gel solidifies and forms a drug reservoir inside the bladder. Upon contact with urine the gel dissolves and is cleared out from the bladder.

Intravesical MMC using TheraCoat gel is expected to increase treatment efficiency due to prolongation of treatment duration and consequently improving bladder exposure to MMC.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Patients with bladder cancer designated to undergo Radical Cystectomy

Exclusion Criteria:

* Sensitivity to MMC
* Acute urinary Tract Infection (UTI)
* Upper urinary tract obstruction.
* Patient received neoadjuvant treatment previous to Radical Cystectomy
* Pregnant women as diagnosed by Beta - HCG, or women that are suspected to be pregnant
* Breastfeeding women

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Assessment of systemic and urine pharmacokinetics of MMC following intravesical instillation of TC-3 mixed with MMC for safety evaluation. | 6 hours
  Study participants undergoing bladder instillation with MMC mixed with TC-3 6 hours prior to radical cystectomy. During these six hours the MMC levels in urine and blood will be measured every hour and the Peak Plasma Concentration (Cmax)and Area under the plasma concentration versus time curve (AUC) will be calculated and compared to the standard toxicity level in patients treated with MMC in saline (standard of cure). In addition, patient tolerability to treatment will be evaluated.

SECONDARY OUTCOMES:
Assessment of the levels of MMC in patients urinary bladder following intravesical instillation of TC-3 mixed with MMC. | 6 hours
  Study participants undergoing bladder instillation with MMC mixed with TC-3 6 hours prior to radical cystectomy. Local (bladder) tissue levels of MMC will be evaluated and compared to MMC levels detected following treatment with MMC in saline (standard of cure).

CONTACTS AND LOCATIONS:
Overall Officials: Michal Jeshurun, MD, Study Director — UroGen Pharma Ltd.
Locations (3):
- Israel (3):
  - Barzilai Hospital, Ashkelon
  - Wolfson, Holon
  - Beilinson, Petah Tikva